CLINICAL TRIAL: NCT01937871
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Parallel-Design, Multicenter Study to Evaluate the Efficacy and Safety of Tadalafil Once-Daily Dosing for 12 Weeks in Men With Signs and Symptoms of Benign Prostatic Hyperplasia and Erectile Dysfunction
Brief Title: A Study of Tadalafil in Men With Benign Prostatic Hyperplasia (BPH) and Erectile Dysfunction (ED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14393; H6D-MC-LVJE (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-09-04; First posted 2013-09-10 (Estimated); Results first posted 2017-02-07 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-05

CONDITIONS: Benign Prostate Hyperplasia; Erectile Dysfunction
MeSH Terms: conditions — Prostatic Hyperplasia; Erectile Dysfunction | interventions — Tadalafil; Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo matching tadalafil or tamsulosin administered once daily by mouth for 16 weeks.
  Interventions: Drug: Placebo
- 5 mg Tadalafil (Experimental): Placebo administered once daily by mouth for 4 weeks during the single-blind placebo run-in period.
  Tadalafil 5 milligram (mg) tablet administered once daily by mouth for 12 weeks during the double-blind treatment period
  Interventions: Drug: 5 mg Tadalafil; Drug: Placebo
- 0.2 mg Tamsulosin (Other): Placebo administered once daily by mouth for 4 weeks during the single-blind placebo run-in period.
  Tamsulosin 0.2 mg capsule administered once daily by mouth for 12 weeks during the double-blind treatment period
  Interventions: Drug: Placebo; Drug: 0.2 mg Tamsulosin

INTERVENTIONS:
Drug: 5 mg Tadalafil — Administered orally
  Other Names: LY450190
  Arms: 5 mg Tadalafil
Drug: Placebo — Administered orally
Drug: 0.2 mg Tamsulosin — Administered orally
  Arms: 0.2 mg Tamsulosin

SUMMARY:
The purpose of this study is to see whether tadalafil can reduce the signs and symptoms in men with Erectile Dysfunction (ED) and Benign Prostatic Hyperplasia-Lower Urinary Tract Symptoms (BPH-LUTS) and improve their quality of life.

ELIGIBILITY:
Main Inclusion Criteria:

* Present with a history of ED and signs and symptoms of BPH.
* Are sexually active with an adult female partner, and expect to remain sexually active with the same adult female partner for the duration of the study.

Main Exclusion Criteria:

* Current treatment with nitrates.
* Prostate-specific antigen (PSA) greater than 10.0 nanogram (ng)/mL at 1st screening.
* PSA greater than or equal to 4.0 to less than or equal to 10.0 ng/mL at 1st screening if prostate malignancy has not been ruled out to the satisfaction of a urologist
* Suffering from other urinary disease like cancer, or infection
* Serious cardiovascular disease
* History of significant renal insufficiency

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 909 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (14):
- China (14):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changchun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changsha
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chengdu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chongqing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hefei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nanchang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nanjing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wenzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wuhan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Xi'an

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.2 mg Tamsulosin: Placebo administered once daily by mouth for 4 weeks during the single-blind placebo run-in period Tamsulosin 0.2 mg capsule administered once daily by mouth for 12 weeks during the double-blind treatment period.
Period: Overall Study
Arm/Group | Placebo | 5 mg Tadalafil | 0.2 mg Tamsulosin
Started | 361 | 363 | 185
Received at Least One Dose of Study Drug | 361 | 362 | 185
Completed | 337 | 346 | 174
Not Completed | 24 | 17 | 11
Not completed — Adverse Event | 6 | 6 | 2
Not completed — Lost to Follow-up | 8 | 2 | 4
Not completed — Withdrawal by Subject | 9 | 6 | 4
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Entry Criteria Not Met | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 5 mg Tadalafil | 0.2 mg Tamsulosin | Total
Number analyzed (Participants) | 361 | 363 | 185 | 909
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (7.35) | 61.8 (7.27) | 61.9 (7.06) | 61.8 (7.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 361 | 363 | 185 | 909
Region of Enrollment [Count of Participants; unit: Participants]
  China | 279 | 277 | 143 | 699
  Korea, Republic of | 71 | 71 | 35 | 177
  Taiwan | 11 | 15 | 7 | 33

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total International Prostate Symptom Score (IPSS) at Week 12
Description: IPSS Total Score is the sum of Questions 1 through 7 of the IPSS questionnaire. Each question was scored from 0 (none/no symptoms) to 5 (frequent symptoms) for an IPSS Total Score ranging from 0 to 35 points; higher numerical scores from the IPSS questionnaire represent greater severity of symptoms. Least squares (LS) mean of change from baseline to endpoint is from an analysis mixed model for repeated measures (MMRM).The model includes effects for treatment, country/region, prior alpha-blocker therapy, baseline Erectile dysfunction (ED) severity (mild/moderate/severe),visit, treatment-by-visit interaction, centered baseline value (defined as the baseline value for a participant - the overall baseline mean value), placebo lead-in total IPSS change (change from Visit 2 at Visit 3), centered baseline-by-treatment.The centered baseline-by-treatment and treatment-by-country interactions was removed if p >= 0.10.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of the study drug, had a baseline and at least one post-baseline IPSS measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 5 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 346 | 354 | 181
units on a scale | -4.08 (0.402) | -5.49 (0.395) | -4.92 (0.493)
Statistical Analysis 1: Comparison: Placebo vs 5 mg Tadalafil; Test type: Superiority or Other; Mean Difference (Final Values) = -1.41, 95% CI 2-sided [-2.25 to -0.57]

2. Secondary Outcome: Change From Baseline in International Index of Erectile Function (IIEF) Erectile Function (EF) Domain at Week 12
Description: IIEF is a 15 item self-reported questionnaire to assess overall erectile function and satisfaction during the past 4 weeks. IIEF- EF is the sum of Questions 1-5 and 15 of the IIEF. Questions 1-5 are scored 0(low/no erectile function) to 5(high erectile function) and Question 15 is scored 1(very low confidence) to 5(very high confidence) with a total score ranging from 1 to 30.Higher scores represent better erectile function.LS mean of change from baseline to endpoint is from MMRM.The model includes effects for treatment,country/region,baseline lower urinary tract symptoms(LUTS) severity (moderate/severe),visit,treatment-by-visit interaction,centered baseline value(defined as the baseline value for a participant-the overall baseline mean value), placebo lead-in total IPSS change(change from Visit 2 at Visit 3),centered baseline-by-treatment and treatment-by-country/region interactions.The centered baseline-by-treatment and treatment-by-country interactions was removed if p >= 0.10.
Time Frame: Baseline, Week 12
Population: All randomized participants who had at least one dose of the study drug, had a baseline and at least one post-baseline IIEF measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 5 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 346 | 354 | 181
units on a scale | 1.88 (0.448) | 5.24 (0.439) | 2.64 (0.556)

3. Secondary Outcome: Change From Baseline in Yes Responses to Question 2 of the Sexual Encounter Profile (SEP) Questionnaire at Week 12
Description: Participant-assessed diary assesses the mean change from baseline in the percentage of "yes" responses to SEP Q2, "Were you able to insert your penis into your partner's vagina?". The SEP Q2 score was determined as the percentage of "yes" responses to SEP Q2 out of all sexual attempts recorded during the time period. Change is defined as the percentage of "yes" responses at endpoint minus the percentage of "yes" responses at baseline. Least squares (LS) mean of change from baseline to endpoint is from an analysis of covariance (ANCOVA). The model includes terms for treatment, country/region, baseline ED severity (mild/moderate/severe), centered baseline value (defined as the baseline value for a participant - the overall baseline mean value), placebo lead-in total IPSS change (change from Visit 2 at Visit 3), the centered baseline-by-treatment and the treatment-by-country/region interactions. The interaction terms are removed if p >= 0.10.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of the study drug, had a baseline and at least one post-baseline SEP measurement. Last Observation Carried Forward (LOCF) was used to impute missing post-baseline values.
Measure: Least Squares Mean (Standard Error); unit: percentage of "yes" responses
Arm/Group | Placebo | 5 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 339 | 350 | 180
percentage of "yes" responses | 10.90 (2.618) | 23.87 (2.548) | 6.84 (3.074)

4. Secondary Outcome: Change From Baseline in Yes Responses to Question 3 of the SEP Questionnaire at Week 12
Description: Participant-assessed diary assesses the mean change from baseline in the percentage of "yes" responses to SEP Q3, "Did your erection last long enough for you to have successful intercourse?".The SEP Q3 score is determined as the percentage of "yes" responses to SEP Q3 out of all sexual attempts recorded during the time period. Change was defined as the percentage of "yes" responses at endpoint minus percentage of "yes" responses at baseline. Least squares (LS) mean of change from baseline to endpoint is from an analysis of covariance (ANCOVA). The model includes terms for treatment, country/region, baseline ED severity (mild/moderate/severe), centered baseline value (defined as the baseline value for a participant - the overall baseline mean value), placebo lead-in total IPSS change (change from Visit 2 at Visit 3), the centered baseline-by-treatment and the treatment-by-country/region interactions. The interaction terms are removed if p >= 0.10.
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage of "yes" responses
Arm/Group | Placebo | 5 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 339 | 350 | 180
percentage of "yes" responses | 15.96 (3.016) | 36.62 (2.935) | 17.42 (3.557)

5. Secondary Outcome: Change From Baseline in IPSS at Week 12
Description: IPSS Total Score is the sum of Questions 1 through 7 of the IPSS questionnaire. Each question is scored from 0 (none/no symptoms) to 5 (frequent symptoms) for an IPSS Total Score ranging from 0 to 35 points; higher numerical scores from the IPSS questionnaire represent greater severity of symptoms. Least squares (LS) mean of change from baseline to endpoint is from an analysis mixed model for repeated measures (MMRM).The model includes effects for treatment, country/region, prior alpha-blocker therapy, baseline Erectile dysfunction (ED) severity (mild/moderate/severe),visit, treatment-by-visit interaction, centered baseline value (defined as the baseline value for a participant - the overall baseline mean value), placebo lead-in total IPSS change (change from Visit 2 at Visit 3), centered baseline-by-treatment. The centered baseline-by-treatment and treatment-by-country interactions was removed if p >= 0.10.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 5 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 346 | 354 | 181
units on a scale | -4.08 (0.402) | -5.49 (0.395) | -4.92 (0.493)
Statistical Analysis 1: Comparison: Placebo vs 0.2 mg Tamsulosin; Test type: Superiority or Other; Mean Difference (Final Values) = -0.85, 95% CI 2-sided [-1.87 to 0.18]

6. Secondary Outcome: Change From Baseline in Uroflowmetry Measures at Week 12
Description: Qmax is defined as the peak urine flow rate (measured in milliliters per second [mL/sec] using standard calibrated flowmeter).
  At each visit, a uroflowmetry assessment was considered valid and the data were included only if the prevoid total bladder volume (assessed by ultrasound) was >=150 to <=550 milliliters (mL) and the voided volume (Vcomp) was >=125 mL. Changes in Qmax from baseline to endpoint in the double-blind treatment period were analyzed using Type III sums of squares ANOVA on rank-transformed data with a term for treatment group.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of the study drug, had a baseline and at least one post-baseline Uroflowmetry measurement.
Measure: Mean (Standard Deviation); unit: Milliliters/seconds (mL/sec)
Groups:
- 5 mg Tadalafil: Placebo administered once daily by mouth for 4 weeks during the single-blind placebo run-in period.Tadalafil 5 milligram (mg) tablet administered once daily by mouth for 12 weeks during the double-blind treatment period.
Arm/Group | Placebo | 5 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 297 | 313 | 154
Milliliters/seconds (mL/sec) | 1.5 (5.46) | 1.9 (5.68) | 2.0 (5.37)

7. Secondary Outcome: Change From Baseline in Postvoid Residual Volume (PVR) at Week 12
Description: The amount of urine remaining in the bladder after void completion.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of the study drug, had a baseline and at least one post-baseline PVR measurement.
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | Placebo | 5 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 341 | 351 | 174
milliliters (mL) | -6.3 (47.86) | -3.8 (49.02) | -9.5 (44.76)

8. Secondary Outcome: Change From Baseline in IPSS Storage (Irritative) Subscore at Week 12
Description: IPSS Storage (Irritative) subscore is the sum of Questions 2, 4 and 7 of the IPSS questionnaire. Scores ranged from 0 (no irritative symptoms) to 5 (frequent irritative symptoms), with total subscore of the 3 questions for irritative subscore ranging from 0 to 15; higher numerical scores from the IPSS questionnaire represent greater severity of symptoms. Least squares (LS) mean of change from baseline to endpoint is from an analysis mixed model for repeated measures (MMRM). The model includes effects for treatment, country/region, prior alpha-blocker therapy, baseline ED severity (mild/moderate/severe), visit, treatment-by-visit interaction, centered baseline value (defined as the baseline value for a participant - the overall baseline mean value), placebo lead-in total IPSS change (change from Visit 2 at Visit 3), centered baseline-by-treatment and treatment-by-country/region interactions.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 5 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 346 | 354 | 181
units on a scale | -1.68 (0.176) | -2.01 (0.173) | -1.90 (0.215)

9. Secondary Outcome: Change From Baseline in IPSS Voiding (Obstructive) Subscore at Week 12
Description: IPSS voiding (obstructive) subscore is the sum of Questions 1, 3, 5 and 6 of the IPSS questionnaire. Scores ranged from 0 (no obstructive symptoms) to 5 (frequent obstructive symptoms), with total subscore of the 4 questions of the obstructive score ranging from 0 to 20; higher numerical scores from the IPSS questionnaire represent greater severity of symptoms. Least squares (LS) mean of change from baseline to endpoint is from an analysis mixed model for repeated measures (MMRM). The model includes effects for treatment, country/region, prior alpha-blocker therapy, baseline ED severity (mild/moderate/severe),visit, treatment-by-visit interaction, centered baseline value (defined as the baseline value for a participant - the overall baseline mean value), placebo lead-in total IPSS change (change from Visit 2 at Visit 3), centered baseline-by-treatment and treatment-by-country/region interactions.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 5 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 346 | 354 | 181
units on a scale | -2.42 (0.271) | -3.49 (0.266) | -3.07 (0.331)

10. Secondary Outcome: Change From Baseline in IPSS Quality of Life (QoL) Index at Week 12
Description: IPSS QoL assess participant response to the following question:"If you were to spend the rest of your life with your urinary condition just the way it is now, how would you feel about that?". Response options are Delighted(0),Pleased(1);Mostly satisfied(2);mixed about equally satisfied and dissatisfied(3);Mostly dissatisfied(4);Unhappy(5);Terrible(6),with a total ranging from 0 to 6; higher numerical scores from the IPSS questionnaire represent greater severity of symptoms. Least squares(LS) mean of change from baseline(bl) to endpoint is from MMRM.The model includes effects for treatment,country/region, prior alpha-blocker therapy,baseline ED severity (mild/moderate/severe),visit, treatment-by-visit interaction, centered bl value (defined as the bl value for a participant -the overall bl mean value),placebo lead-in total IPSS change(change from Visit 2 at Visit 3),centered bl-by-treatment and treatment-by-country/region interactions.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of the study drug, had a baseline and at least one post-baseline QoL measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 5 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 346 | 354 | 181
units on a scale | -0.85 (0.099) | -0.98 (0.097) | -1.00 (0.121)

11. Secondary Outcome: Number of Participants With Patient Global Impression of Improvement (PGI-I) at Week 12
Description: PGI-I measures a participant's perception of improvement at the time of assessment compared with the start of treatment. Score ranges from 1 (very much better) to 7 (very much worse).
Time Frame: Week 12
Population: All randomized participants who received at least one dose of the study drug, had a baseline and at least one post-baseline PGI-I measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 5 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 342 | 353 | 176
Participants
  Very Much Worse | 0 | 0 | 0
  Much Worse | 3 | 2 | 0
  A Little Worse | 5 | 2 | 1
  No Change | 87 | 53 | 37
  A Little Better | 169 | 164 | 93
  Much Better | 73 | 119 | 39
  Very Much Better | 5 | 13 | 6

12. Secondary Outcome: Number of Participants With Clinician Global Impression of Improvement (CGI-I) at Week 12
Description: CGI-I measures clinician's perception of participant improvement at the time of assessment (compared with the start of treatment) with scores ranging from 1 (very much better) to 7 (very much worse).
Time Frame: Week 12
Population: All randomized participants who received at least one dose of the study drug and had a baseline and at least one post-baseline CGI-I measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 5 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 343 | 353 | 176
Participants
  Very Much Worse | 0 | 1 | 0
  Much Worse | 2 | 0 | 0
  A Little Worse | 12 | 5 | 1
  No Change | 91 | 66 | 39
  A Little Better | 130 | 140 | 85
  Much Better | 92 | 120 | 41
  Very Much Better | 16 | 21 | 10

13. Secondary Outcome: Change From Baseline in IIEF Overall Satisfaction (OS) at Week 12
Description: IIEF is a 15 item self-reported questionnaire used to assess overall erectile function and satisfaction during the past 4 weeks. IIEF-OS is the sum of Questions 13 and 14. Scores range from 1 (low/no satisfaction) to 5 (high satisfaction) for each question, with a total subscore ranging from 2 to 10;higher scores represent better erectile function. Least squares (LS) mean of change from baseline to endpoint is from an analysis mixed model for repeated measures (MMRM). The model includes effects for treatment, country/region, baseline LUTS severity (moderate/severe), visit, treatment-by-visit interaction,centered baseline value (defined as the baseline value for a participant - the overall baseline mean value), placebo lead-in total IPSS change (change from Visit 2 at Visit 3), centered baseline-by-treatment and treatment-by-country/region interactions. The centered baseline-by-treatment and treatment-by-country interactions was removed if p >= 0.10.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of the study drug, had a baseline and at least one post-baseline IIEF measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 5 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 346 | 354 | 181
units on a scale | 0.62 (0.120) | 1.54 (0.118) | 0.71 (0.150)

14. Secondary Outcome: Change From Baseline in IIEF Intercourse Satisfaction at Week 12
Description: IIEF is a 15 item self-reported questionnaire used to assess overall erectile function and satisfaction during the past 4 weeks. IIEF-IS is the sum of Questions 6,7 and 8 of the IIEF. Scores range from 0(low/no satisfaction) to 5(high satisfaction) for each question, with the total possible score for the 3 questions ranging from 0 to 15.Higher scores were indicative of an increase in intercourse satisfaction. Least squares (LS) mean of change from baseline to endpoint is from MMRM. The model includes effects for treatment, country/region, baseline LUTS severity (moderate/severe), visit, treatment-by-visit interaction,centered baseline value(defined as the baseline value for a participant- the overall baseline mean value), placebo lead-in total IPSS change (change from Visit 2 at Visit 3), centered baseline-by-treatment and treatment-by-country/region interactions. The centered baseline-by-treatment and treatment-by-country interactions was removed if p >= 0.10.
Time Frame: Baseline, Week 12
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 5 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 346 | 354 | 181
units on a scale | -0.05 (0.183) | 1.08 (0.179) | 0.41 (0.227)

15. Secondary Outcome: Change From Baseline in IIEF Orgasmic Function at Week 12
Description: IIEF is a 15 item self-reported questionnaire used to assess overall erectile function and satisfaction during the past 4 weeks. IIEF orgasmic function is the sum of Q9 and Q10 of the IIEF. Scores ranged from 0 (no stimulation) to 5 (almost always) for each question, with the total possible score for the 2 questions ranging from 0 to 10. Higher scores were indicative of better orgasmic function. Least squares (LS) mean of change from baseline to endpoint is from MMRM. The model includes effects for treatment, country/region, baseline LUTS severity (moderate/severe), visit, treatment-by-visit interaction, centered baseline value (defined as the baseline value for a participant - the overall baseline mean value), placebo lead-in total IPSS change (change from Visit 2 at Visit 3), centered baseline-by-treatment and treatment-by-country/region interactions. The centered baseline-by-treatment and treatment-by-country interactions was removed if p >= 0.10.
Time Frame: Baseline, Week 12
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 5 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 346 | 354 | 181
units on a scale | 0.28 (0.169) | 1.31 (0.165) | 0.57 (0.207)

16. Secondary Outcome: Change From Baseline in IIEF Sexual Desire at Week 12
Description: IIEF is a 15 item self-reported questionnaire used to assess overall erectile function and satisfaction during the past 4 weeks. IIEF sexual desire is the sum of Q11 and Q12. Scores ranged from 1 (low/almost never) to 5 (very high/almost always) for each question, with the total possible score for the 2 questions ranging from 2 to 10. Higher scores were indicative of increased sexual desire. Least squares (LS) mean of change from baseline to endpoint is from MMRM. The model includes effects for treatment, country/region, baseline LUTS severity (moderate/severe), visit, treatment-by-visit interaction, centered baseline value (defined as the baseline value for a participant - the overall baseline mean value), placebo lead-in total IPSS change (change from Visit 2 at Visit 3), centered baseline-by-treatment and treatment-by-country/region interactions. The centered baseline-by-treatment and treatment-by-country interactions was removed if p >= 0.10.
Time Frame: Baseline, Week 12
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 5 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 346 | 354 | 181
units on a scale | 0.46 (0.114) | 1.12 (0.111) | 0.28 (0.142)

17. Secondary Outcome: Change From Baseline in IIEF Subscores at Week 12
Description: IIEF Question 3 asks how often a participant was able to penetrate his partner over the past 4 weeks. Scores range from 0 (did not attempt intercourse) to 5 (almost always or always). IIEF Question 4 asks whether/how often a participant was able to maintain an erection after penetration over the past 4 weeks. Scores range from 0 (did not attempt intercourse) to 5 (almost always or always). Least squares (LS) mean of change from baseline to endpoint is from MMRM. The model includes effects for treatment, country/region, baseline LUTS severity (moderate/severe), visit, treatment-by-visit interaction, centered baseline value (defined as the baseline value for a participant - the overall baseline mean value), placebo lead-in total IPSS change (change from Visit 2 at Visit 3), centered baseline-by-treatment and treatment-by-country/region interactions. The centered baseline-by-treatment and treatment-by-country interactions was removed if p >= 0.10.
Time Frame: Baseline, Week 12
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 5 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 346 | 354 | 181
units on a scale
  IIEF Question 3 | 0.28 (0.097) | 0.87 (0.095) | 0.39 (0.120)
  IIEF Question 4 | 0.30 (0.093) | 0.87 (0.091) | 0.50 (0.115)

18. Secondary Outcome: Change From Baseline in Total IPSS at Week 4 and Week 8
Description: IPSS Total Score is the sum of Questions 1 through 7 of the IPSS questionnaire. Each question is scored from 0 (none/no symptoms) to 5 (frequent symptoms) for an IPSS Total Score ranging from 0 to 35 points; higher numerical scores from the IPSS questionnaire represent greater severity of symptoms. Least squares (LS) mean of change from baseline to endpoint is from an analysis mixed model for repeated measures (MMRM). The model includes effects for treatment, country/region, prior alpha-blocker therapy, baseline ED severity (mild/moderate/severe),visit, treatment-by-visit interaction, centered baseline value (defined as the baseline value for a participant - the overall baseline mean value), placebo lead-in total IPSS change (change from Visit 2 at Visit 3), centered baseline-by-treatment. The centered baseline-by-treatment and treatment-by-country interactions was removed if p >= 0.10.
Time Frame: Baseline, Week 4; Baseline, Week 8
Population: All randomized participants who had at least one dose of the study, had a baseline and at least one post-baseline IPSS measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 5 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 346 | 354 | 181
units on a scale
  Week 4 | -2.99 (0.365) | -4.10 (0.359) | -3.92 (0.434)
  Week 8 | -3.50 (0.385) | -4.85 (0.378) | -4.44 (0.465)

19. Secondary Outcome: Change From Baseline in IIEF EF at Week 4 and Week 8
Description: IIEF is a 15 item self-reported questionnaire used to assess overall erectile function and satisfaction during the past 4 weeks. IIEF- EF is the sum of Questions 1-5 and 15 of the IIEF. Questions 1-5 were scored 0 (low/no erectile function) to 5 (high erectile function) and Question 15 was scored 1 (very low confidence) to 5 (very high confidence) with a total score ranging from 1 to 30. Higher scores represent better erectile function. LS mean of change from baseline to endpoint is from MMRM. The model includes effects for treatment, country/region, baseline LUTS severity (moderate/severe), visit, treatment-by-visit interaction, centered baseline value (defined as the baseline value for a participant - the overall baseline mean value), placebo lead-in total IPSS change (change from Visit 2 at Visit 3), centered baseline-by-treatment and treatment-by-country/region interactions. The centered baseline-by-treatment and treatment-by-country interactions was removed if p >= 0.10.
Time Frame: Baseline, Week 4; Baseline, Week 8
Population: All randomized participants who had at least one dose of the study, had a baseline and at least one post-baseline IIEF measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 5 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 346 | 354 | 181
units on a scale
  Week 4 | 1.23 (0.412) | 4.50 (0.403) | 1.43 (0.498)
  Week 8 | 1.51 (0.423) | 4.77 (0.414) | 2.19 (0.516)

20. Secondary Outcome: Change From Baseline in Yes Responses to Question 2 of the SEP Questionnaire at Week 4 and Week 8
Description: Participant-assessed diary assesses the mean change from baseline in the percentage of "yes" responses to SEP Q2, "Were you able to insert your penis into your partner's vagina?". The SEP Q2 score is determined as the percentage of "yes" responses to SEP Q2 out of all sexual attempts recorded during the time period. Change was defined as the percentage of "yes" responses at endpoint minus the percentage of "yes" responses at baseline. Least squares (LS) mean of change from baseline to endpoint is from an analysis of covariance (ANCOVA). The model includes terms for treatment, country/region, baseline ED severity (mild/moderate/severe), centered baseline value (defined as the baseline value for a participant - the overall baseline mean value), placebo lead-in total IPSS change (change from Visit 2 at Visit 3), the centered baseline-by-treatment and the treatment-by-country/region interactions. The interaction terms are removed if p >= 0.10.
Time Frame: Baseline, Week 4; Baseline, Week 8
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage of "yes" responses
Arm/Group | Placebo | 5 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 338 | 350 | 179
percentage of "yes" responses
  Week 4: number analyzed (Participants) | 328 | 344 | 175
  Week 4 | 5.43 (2.394) | 20.53 (2.325) | 6.21 (2.827)
  Week 8 | 10.79 (2.510) | 23.22 (2.441) | 7.42 (2.950)

21. Secondary Outcome: Change From Baseline in Yes Responses to Question 3 of the SEP Questionnaire at Week 4 and Week 8
Description: Participant-assessed diary assesses the mean change from baseline in the percentage of "yes" responses to SEP Q3, "Did your erection last long enough for you to have successful intercourse?". The SEP Q3 score is determined as the percentage of "yes" responses to SEP Q3 out of all sexual attempts recorded during the time period. Change was defined as the percentage of "yes" responses at endpoint minus percentage of "yes" responses at baseline. Least squares (LS) mean of change from baseline to endpoint is from an analysis of covariance (ANCOVA). The model includes terms for treatment, country/region, baseline ED severity (mild/moderate/severe), centered baseline value (defined as the baseline value for a participant - the overall baseline mean value), placebo lead-in total IPSS change (change from Visit 2 at Visit 3), the centered baseline-by-treatment and the treatment-by-country/region interactions. The interaction terms are removed if p >= 0.10.
Time Frame: Baseline, Week 4; Baseline, Week 8
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage of "yes" responses
Arm/Group | Placebo | 5 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 338 | 350 | 179
percentage of "yes" responses
  Week 4: number analyzed (Participants) | 328 | 344 | 175
  Week 4 | 7.41 (2.701) | 23.38 (2.622) | 9.57 (3.213)
  Week 8 | 14.08 (2.884) | 32.27 (2.805) | 14.98 (3.411)

22. Secondary Outcome: Change From Baseline in Modified International Prostate Symptom Score (mIPSS) at Week 2
Description: The modified IPSS is the total IPSS collected at 2 weeks post-baseline.The total IPSS is obtained by combining the scores of the responses to component questions 1 through 7. Each question is scored from 0-5 for a total IPSS range of 0-35 points; higher numerical scores from the IPSS questionnaire represent greater severity of symptoms. Least squares (LS) mean of change from baseline to endpoint is from ANCOVA. The model includes terms for treatment, country/region, prior alpha-blocker use and baseline ED severity (mild/moderate/severe), centered baseline value (defined as the baseline value for a participant - the overall baseline mean value), placebo lead-in total IPSS change (change from Visit 2 at Visit 3), the centered baseline-by-treatment and the treatment-by-country/region interactions. The interaction terms are removed if p >= 0.10.
Time Frame: Baseline, Week 2
Population: All randomized participants who received at least one dose of the study drug, had a baseline and at least one post-baseline mIPSS measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 5 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 352 | 358 | 183
units on a scale | -2.19 (0.342) | -3.40 (0.336) | -3.20 (0.403)

ADVERSE EVENTS:
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | Placebo | 5 mg Tadalafil | 0.2 mg Tamsulosin
Serious Adverse Events (participants affected / at risk) | 5/361 | 7/362 | 2/185
Other Adverse Events (participants affected / at risk) | 62/361 | 64/362 | 21/185
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=361) | 5 mg Tadalafil (N=362) | 0.2 mg Tamsulosin (N=185)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Melanosis coli (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=361) | 5 mg Tadalafil (N=362) | 0.2 mg Tamsulosin (N=185)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Type v hyperlipidaemia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Refraction disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal mass (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Gastrointestinal hypermotility (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Hyperchlorhydria (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal cyst (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Body tinea (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (5) | 8 (8) | 2 (2)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 4 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 3 (3) | 5 (5) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood urine (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood urine present (Investigations) | 2 (2) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (6) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (3) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 6 (6) | 3 (3) | 5 (5)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Enuresis (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Prostatic calcification (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pemphigus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days